CLINICAL TRIAL: NCT03509077
Title: Study of Addiction Criteria in the Elderly
Acronym: CAPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0046; 2018-A00905-50 (Other: ID-RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-04-26 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Depressive Disorder
Keywords: geriatric; addiction
MeSH Terms: conditions — Depressive Disorder; Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients over 65 years old who are exposed to alcohol or benzodiazepines will be recruited through the Fragility Assessment and Addictions Prevention Day Hospital, the Addiction Service and the Geriatric Post-Emergency Department. Toulouse University Hospital.

The investigators will study descriptively the frequency of substance use disorder and the frequency of DSM-5 criteria associated with this diagnosis in a population of elderly subjects.

DETAILED DESCRIPTION:
The hypothesis of this research is that some of the DSM-5 criteria for substance use disorder are more appropriate than others in people over 65 years of age. This study therefore aims to describe the frequency of the DSM-5 criteria for the substance use disorder in a population over 65 years of age and to link it secondarily to the severity of the addiction.

The study is a descriptive study of a population of subjects over 65 years old. It aims to search for addiction criteria in this population by formulating the hypothesis of an addictive vulnerability relating to certain risk factors.

To sensitize the detection of criteria, we chose among older subjects those who are most at risk because they are more exposed to the vulnerability factor relative to this population (physical disability, loss of autonomy, loneliness).

ELIGIBILITY:
Inclusion Criteria:

* To be over 65
* Have given your non-oral opposition to participate in research
* Mini-Mental State Examination (MMSE) greater than or equal to 24
* Be part of one of the 3 inclusion services of the University Hospital of Toulouse
* For 12 months, have daily consumption of benzodiazepine (at least once a day) and / or have excessive alcohol consumption as recommended by the American Geriatric Society (more than one unit of alcohol per day) ).

Exclusion Criteria:

* Patient refusing to participate in the study
* MMSE less than 24
* Acute decompensation of a psychiatric disorder
* Impossibility to understand or speak French
* Patient under the protection of justice

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Three groups of patients will be recruited in three departments of the University Hospital of Toulouse:
  1. Patients meeting the criteria for frailty will be recruited to the Fragility Assessment and Addiction Prevention Day Hospital.
  2. Patients over 65, addicts and consultant in a specialized service.
  3. Patients who have decompensated their fragility criteria will be recruited from the geriatric post-emergency department of Toulouse University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-06-19 (Estimated); Study Completion 2019-06-19 (Estimated)

PRIMARY OUTCOMES:
The number of DSM-5 criteria | 1 hour
  The number of DSM-5 criteria for substance use disorder in the patient assessment.
  The number of DSM-5 criteria is a method of problematic substance use leading to clinically significant impairment or impairment characterized by the presence of at least two of the following manifestations over a 12-month period

SECONDARY OUTCOMES:
The Mini-GDS : a screening tool | 1 hour
  The diagnosis of depression will be made using a screening tool, the Mini-GDS, performed in routine clinical practice as part of the assessment at the day hospital for frailty and addiction prevention.
  The Mini-GDS includes 4 items rated at one point depending on the answer. A higher score 1 makes it possible to suspect the existence of a depression.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Salles, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No